CLINICAL TRIAL: NCT07165197
Title: Visual Performance of Clareon® Vivity® and PureSee® Intraocular Lenses in Patients Undergoing Cataract Surgery
Brief Title: Visual Performance of Clareon Vivity and PureSee IOL
Acronym: PURVI2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OMIQ Research (Network)
Responsible Party: Principal Investigator, Merce Guarro, MD, OMIQ Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOR2025-HGC-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended depth of focus intraocular lens Clareon Vivity (Experimental)
  Interventions: Device: Phacoemulsification with implantation of an extended depth of focus intraocular lens
- Extended depth of focus intraocular lens PureSee (Active Comparator)
  Interventions: Device: Phacoemulsification with implantation of an extended depth of focus intraocular lens

INTERVENTIONS:
Device: Phacoemulsification with implantation of an extended depth of focus intraocular lens — Comparison of two different Extended depth of focus intraocular lenses

SUMMARY:
This is study to determine the visual performance of patients with age-related cataracts implanted in both eyes with either of two extended depth of focus intraocular lenses, the Clareon Vivity (Alcon Healthcare) or the PureSee (Johnson & Johnson)

ELIGIBILITY:
Inclusion Criteria:

* Patients of any sex and race aged 50 years or older
* Patients undergoing bilateral age-related cataract surgery with a lens opacity grade 3 or higher in the LOCS III grading scale
* Willing to receive implantation of an EDOF IOL
* Willing to sign the informed consent and attend the study visits

Exclusion Criteria:

* Requirement of a spherical or toric power of the IOL to achieve emmetropia beyond the available range of either of the two lenses
* The number of patients included with low astigmatism that require an equivalent to a T2 toric IOL will be capped to 10 patients/group
* Irregular astigmatism
* Contact lens wear in the previous 3 weeks before biometry
* Moderate or severe ocular surface, corneal, macular or optic nerve disease that in opinion of the investigator precludes the desired functional results
* History of previous refractive, cornea, retina or glaucoma surgery
* Eyes with a clear lens demanding a refractive lens exchange
* Amblyopia in any eye
* Significant previous ocular trauma
* Pregnancy
* A systemic condition that, in the opinion of the investigator, precludes the reliable assessments required in the study (i.e., dementia) or participation in the study (i.e., severe mobility problems).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Distance-corrected binocular defocus curve at 4 m | 3 months

SECONDARY OUTCOMES:
Monocular and binocular, corrected and uncorrected distance, intermediate, and near visual acuities | 3 months
  Visual acuities in logMAR scale using ETDRS (Early Treatment Diabetic Retinopathy Study) charts
Distance-corrected contrast sensitivity | Three months
  Contrast sensitivity using M&S device
Low contrast (25%) binocular distance-corrected visual acuity | 3 months
  Contrast sensitivity in logMAR scale using low contrast ETDRS (Early Treatment Diabetic Retinopathy Study) charts
Visual dysfunction assessment using the QUVID (Questionnaire for visual disturbances) questionnaire | 3 months
  Assessment of qualitative visual dysphotopsia using a specific validated questionnaire
Spectacle independence assessment using the IOLSAT (Intraocular lens satisfaction) questionnaire | 3 months
  Assessment of recent use of spectacles to see at different distances using a specific questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- OMIQ Research, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided